CLINICAL TRIAL: NCT00035984
Title: A Phase 3, Randomized, Triple-Blind, Parallel-Group, Long-Term, Placebo-Controlled, Multicenter Study to Examine the Effect on Glucose Control (HbA1c) of AC2993 Given Twice Daily in Subjects With Type 2 Diabetes Mellitus Treated With Metformin and a Sulfonylurea
Brief Title: Evaluation of the Effect on Glucose Control of AC2993 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2993-115
Record Dates: First submitted 2002-05-07; First posted 2002-05-08 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-01

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Type 2 Diabetes Mellitis
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AC2993 5 mcg (0.02 mL) (Experimental): Placebo, then AC2993 5 mcg, then AC2993 5 mcg
  Interventions: Drug: AC2993
- AC2993 10mcg (0.04 mL) (Experimental): Placebo, then AC2993 5 mcg, then AC2993 10 mcg
  Interventions: Drug: AC2993
- Placebo 0.02 mL (Placebo Comparator): Placebo 0.02 mL, then Placebo 0.02 mL, then Placebo 0.02 mL
  Interventions: Drug: Placebo
- Placebo 0.04 mL (Placebo Comparator): Placebo 0.02 mL, then Placebo 0.02 mL, then Placebo 0.04 mL
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AC2993 — Placebo Lead In (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 26 weeks - All are subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 5 mcg (0.02 mL)
Drug: AC2993 — Placebo Lead In (0.02 mL) for 4 weeks / AC2993 5 mcg (0.02 mL) for 4 weeks / AC2993 10 mcg (0.04 mL) for 26 weeks - All are subcutaneously injected twice daily
  Other Names: synthetic exendin-4
  Arms: AC2993 10mcg (0.04 mL)
Drug: Placebo — Placebo Lead In (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 4 weeks / AC2993 5mcg (0.02 mL) for 26 weeks - All are subcutaneously injected twice daily
  Arms: Placebo 0.02 mL
Drug: Placebo — Placebo Lead In (0.02 mL) for 4 weeks / Placebo mcg (0.02 mL) for 4 weeks / Placebo (0.04 mL) for 26 weeks - All are subcutaneously injected twice daily
  Arms: Placebo 0.04 mL

SUMMARY:
This is a multicenter, randomized, blinded, placebo-controlled study to assess the effects on glucose control of AC2993 as compared to placebo in patients with type 2 diabetes. Patients will be randomized into one of two AC2993 treatment arms or to placebo treatment and will continue with their required existing diabetes medications (metformin and a sulfonylurea) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 2 diabetes mellitus
* Treated with both metformin and a sulfonylurea at defined doses for at least 3 months prior to screening
* BMI= 27-45 kg/m2
* HbA1c value between 7.5% and 11%

Exclusion Criteria:

* Treated with oral anti-diabetic medications other than metformin and sulfonylurea within 3 months of screening
* Patients treated previously with AC2993
* Patients presently treated with insulin

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 734 (Actual)
Dates: Start 2002-05; Primary Completion 2003-08 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c from Baseline to Week 30 | Baseline (Day 1) to Week 30
  Change in HbA1c from Baseline (Day 1) to study termination (Week 30)

SECONDARY OUTCOMES:
Change in HbA1c from baseline (Day 1) to each of the intermediate visits | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24
  Change in HbA1c from baseline, measured from Visit 3 (Day 1) to each of the intermediate visits (Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, and Week 24)
The number of subjects achieving HbA1c target values of < 7% and < 8% by Week 30 | Baseline (Day 1) and Week 30
  The number of subjects achieving HbA1c target values of < 7% and < 8% by study termination (Week 30)
The number of subjects achieving HbA1c reductions of > 0.5% and > 1.0% by Week 30 | Baseline (Day 1), and Week 30
  The number of subjects achieving HbA1c reductions of > 0.5% and > 1.0% by study termination (Week 30)
The time to achieve specific HbA1c target values of < 7% and < 8% | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24, Week 30
  The time it takes subjects to achieve HbA1c target values of < 7% and < 8%
The time to achieve HbA1c reductions of 0.5% or more and >1.0% or more | Baseline (Day 1), Week 2, Week 4, Week 6, Week 12, Week 18, Week 24, Week 30
  The time it takes subjects to achieve HbA1c reductions of 0.5% or more and >1.0% or more
Change in body weight from Baseline to each intermediate visit and Week 30 | Baseline (Day 1), Week 2, Week 4, Week, 6, Week 12, Week 18, Week 24, Week 30
  Change in body weight (kg) from Baseline to each intermediate visit and Week 30

CONTACTS AND LOCATIONS:
Locations (100):
- United States (100):
  - Pinnacle Research Group, Anniston, Alabama
  - Parkway Medical Center, Birmingham, Alabama
  - Extended Arm Physicians/ Southern Drug, Montgomery, Alabama
  - Southern Drug Research Network, Tallassee, Alabama
  - First Care Family Doctors, Fayetteville, Arkansas
  - Physicians Group Research Clinic, LLC, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - East Bay Clinical Trial Center, Concord, California
  - Medical Group of Encino, Encino, California
  - Valley Research, Fresno, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - Whittier Institute for Diabetes, La Jolla, California
  - Richard Cherlin, M.D., Los Gatos, California
  - Dr. Martinez Medical Clinic, Moreno Valley, California
  - Comprehensive Diabetes-Endocrine Medical Associates, Redwood City, California
  - Radiant Research-San Diego, San Diego, California
  - Veterans Medical Research Foundation, San Diego, California
  - Diablo Clinical Research, Walnut Creek, California
  - Creekside Endocrine Associates, Denver, Colorado
  - University of Colorado-Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - Medstar Clinical Research, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Medical Research Unlimited, Aventura, Florida
  - Morton Plant Mease Health Care, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Internal Medicine Associates, Fort Myers, Florida
  - Clin Sci International, Gainesville, Florida
  - Northeast Florida Endocrine & Diabetes Research, Jacksonville, Florida
  - Jupiter Research Institute, Jupiter, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Comprehensive NeuroScience Inc., Sarasota, Florida
  - Tallahassee Endocrine Associates, Tallahassee, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Columbus Metabolic Foundation, Columbus, Georgia
  - University of Hawaii-Diabetes Research Group, ‘Ewa Beach, Hawaii
  - University Primary Care Center at Belvidere, Belvidere, Illinois
  - Northwestern Memorial Physicians Group, Chicago, Illinois
  - Illinois Center for Clinical Trials, Chicago, Illinois
  - Cook County Hospital, Chicago, Illinois
  - American Health Network, Indianapolis, Indiana
  - Indiana University Outpatient Clinical Research, Indianapolis, Indiana
  - Lipid, Atherosclerosis & Metabolic Clinic, Kansas City, Kansas
  - Kentucky Diabetes Center, Lexington, Kentucky
  - Central Kentucky Research Associates, Lexington, Kentucky
  - University of Kentucky Metabolic Research Group, Lexington, Kentucky
  - MedResearch, Inc., Louisville, Kentucky
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Ochsner Clinic, New Orleans, Louisiana
  - University of Maryland-Joslin Diabetes Center, Baltimore, Maryland
  - Clinica Research Inc., Waltham, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Grand Rapids Associated Interns, Grand Rapids, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Diabetes and Endocrinology Specialists, Chesterfield, Missouri
  - Midwest Pharmaceutical Research, City of Saint Peters, Missouri
  - Medical Arts Research Collaborative, Excelsior Springs, Missouri
  - St Lukes Lipid and Diabetes Research Center, Kansas City, Missouri
  - Mid Missouri Research Specialists, Inc., Rolla, Missouri
  - Radiant Research-St. Louis, St Louis, Missouri
  - Mercury Street Medical, Butte, Montana
  - Lovelace Scientific Resources-Las Vegas, Las Vegas, Nevada
  - Lisa Abbott, MD, Reno, Nevada
  - SUNY Downstate, Brooklyn, New York
  - St. Lukes Roosevelt Hospital, New York, New York
  - Rochester Clinical Research, Rochester, New York
  - DOCS at Beth Israel Medical Center, Yonkers, New York
  - Charlotte Clinical Research, Charlotte, North Carolina
  - UNC Diabetes Care Center, Durham, North Carolina
  - Unifour Medical Research, Hickory, North Carolina
  - New Hanover Medical Research Associates, Wilmington, North Carolina
  - Radiant Research-Columbus, Columbus, Ohio
  - University Mednet, Mentor, Ohio
  - OU Health Sciences Center, Oklahoma City, Oklahoma
  - Medford Medical Clinic, Medford, Oregon
  - Radiant Research, Portland, Oregon
  - Physicians for Clinical Research, Camp Hill, Pennsylvania
  - Thomas Jefferson University Diabetes Research Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Philadelphia Health Associates, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CNS Clinical Trials, Chester, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Holston Medical Group, Kingsport, Tennessee
  - The Endocrine Clinic, Memphis, Tennessee
  - Mid State Endocrine Associates, Nashville, Tennessee
  - Israel A. Hartman, M.D., Arlington, Texas
  - Dallas Diabetes and Endocrinology Research Center, Dallas, Texas
  - Texas Tech University Health Sciences-Internal Medicine, El Paso, Texas
  - North Texas Clinical Research, Irving, Texas
  - University of Texas Health Sciences Center-Texas Diabetes Institute, San Antonio, Texas
  - Diabetes and Glandular Disease Clinic, San Antonio, Texas
  - SAM Clinical Research, San Antonio, Texas
  - Utah Diabetes Center at the University of Utah, Salt Lake City, Utah
  - Salt Lake Research, Salt Lake City, Utah
  - Medical Associates of Northern Virginia, Arlington, Virginia
  - West Olympia Internal Medicine, Olympia, Washington
  - Rockwood Clinic, Spokane, Washington
  - University of Wisconsin West Clinic, Madison, Wisconsin
  - Midwest Endocrinology Associates, Milwaukee, Wisconsin

REFERENCES:
- [Result] Kendall DM, Riddle MC, Rosenstock J, Zhuang D, Kim DD, Fineman MS, Baron AD. Effects of exenatide (exendin-4) on glycemic control over 30 weeks in patients with type 2 diabetes treated with metformin and a sulfonylurea. Diabetes Care. 2005 May;28(5):1083-91. doi: 10.2337/diacare.28.5.1083. PMID 15855571
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356